CLINICAL TRIAL: NCT01730781
Title: Characterization of CB1 Receptors Using [11-C]OMAR
Brief Title: Imaging Cannabinoid Receptors Using Positron Emission Tomography (PET) Scanning
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Deepak C. D'Souza, Associate Professor, Yale University
Other Study IDs: 1005006735; 1R21DA030702-01A1 (NIH); 1R21MH094961-01A1 (NIH)
Record Dates: First submitted 2012-06-14; First posted 2012-11-21 (Estimated); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Schizophrenia; Cannabis Dependence; Prodromal for Psychotic Illness; Family History of Alcoholism; Healthy Control; Opioid-use Disorder; Post Traumatic Stress Disorder
Keywords: Cannabis dependence; Brain Imaging; Schizophrenia; Control; PTSD; OUD
MeSH Terms: conditions — Schizophrenia; Marijuana Abuse; Opioid-Related Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — At the screening visit, genomic DNA will be extracted from whole blood, assigned a code, and stored for analysis of group differences in the frequency of CB1R alleles and to examine the relationship between allelic variation at the CB1R locus and [11-C] OMAR binding. In addition, other genes or markers that may be related to brain function or to behavior may be studied.

GROUPS / COHORTS (7):
- Schizophrenia: Patients diagnosed with schizophrenia both on medication and off medication
  Interventions: Radiation: [11-C]OMAR
- Cannabis dependence: Frequent users of cannabis
  Interventions: Radiation: [11-C]OMAR
- Family history of alcoholism: Healthy volunteers with a first degree relative with alcoholism
  Interventions: Radiation: [11-C]OMAR
- Prodrome for psychotic illness: Not meeting full criteria for psychotic illness but exhibiting prodromal symptoms
  Interventions: Radiation: [11-C]OMAR
- Healthy Volunteers: Healthy volunteers with no current or past major medical or psychiatric history
  Interventions: Radiation: [11-C]OMAR
- PTSD-Post Traumatic Stress Disorder: Patients diagnosed with Post Traumatic Stress Disorder
  Interventions: Radiation: [11-C]OMAR
- Opioid Use Disorder: Patients diagnosed with Opioid Use Disorder
  Interventions: Radiation: [11-C]OMAR

INTERVENTIONS:
Radiation: [11-C]OMAR — The radiotracer, [11-C]OMAR will be administered at no more than 10 micrograms at the beginning of each PET scan.

SUMMARY:
The aim of the present study is to assess the availability of cannabinoid receptors (CB1R) in the human brain. CB1R are present in everyone's brain, regardless of whether or not someone has used cannabis. The investigators will image brain cannabinoid receptors using Positron Emission Tomography (PET) imaging and the radioligand OMAR, in healthy individuals and several conditions including 1) cannabis use disorders, 2) psychotic disorders, 3) prodrome of psychotic illness and 4) individuals with a family history of alcoholism, 5) Post-Traumatic Stress Disorder 6) Opioid Use Disorder using the PET imaging agent or radiotracer, [11C]OMAR. This will allow us to characterize the number and distribution of CB1R in these conditions. It is likely that the list of conditions will be expanded after the collection of pilot data and as new data on cannabinoids receptor function and psychiatric disorders becomes available.

Those in the cannabis us disorder arm of the study will have a PET scan on at least three occasions: once while smoking as usual, once after 48-hours of abstinence from cannabis, and a final time after 4 weeks of abstinence. Additional scans may be conducted within the 4 weeks and the last scan may be conducted well beyond 4 weeks. Similarly, while most schizophrenia patients may get scanned just once, a subgroup of patients may get scanned more than once. For example to tease out the effects of medications, unmedicated patients may get scanned while unmedicated and again after treatment with antipsychotic medications. Similarly prodromes may get scanned while in the prodromal stage off medications, on medications and after conversion to schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Males ages 18-55
* For cannabis users:
* Willing to abstain from cannabis use for four weeks
* For schizophrenia:
* Meets DSM-IV-TR criteria for schizophrenia or schizoaffective disorder
* For prodrome for psychotic illness:
* Meets SIPS criteria for prodromal syndrome
* For family history positive:
* First degree relative with alcoholism
* For Post-Traumatic Stress Disorder
* Meets DSM-IV-TR criteria for PTSD
* For OUD
* Meets DSM-IV-TR criteria for Opioid Use Disorder

Exclusion Criteria:

* Current neuro-psychiatric illness (including cannabis dependence) or severe systemic disease. Cannabis use disorder is permitted in the cannabis dependent group. Schizophrenia and schizoaffective disorder is permitted in the schizophrenia group. Psychotic symptoms are permitted in the prodromal group. Post-Traumatic Stress Disorder is permitted in the PTSD group and Opioid Use Disorder is permitted in the OUD group.
* Presence of ferromagnetic metal in the body or heart pacemaker
* Have had exposure to ionizing radiation that in combination with the study tracer would result in a cumulative exposure that exceeds recommended exposure limits
* Are claustrophobic

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population is composed of schizophrenia, cannabis dependence, prodromal for psychotic illness, family history of alcoholism, healthy volunteers, Post-Traumatic Stress Disorder and Opioid Use Disorder.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-07; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
PET Imaging | One time within 4 weeks of screening
  This study will utilize the radioligand [11C]OMAR and High Resolution Research Tomography (HRRT) Positron Emission Tomography (PET) to measure brain CB1 receptor availability in all study populations.
  Those in the cannabis dependent population of the study will have PET scanning on three occasions: once within four weeks of screening while smoking as usual, once 48-hours later after remaining abstinent, and once four weeks later after remaining abstinent. The change in receptor density at each time point will be evaluated.
  Those in the other populations will have PET scanning done on one occasion within four weeks of screening.

CONTACTS AND LOCATIONS:
Overall Officials: Deepak C D'Souza, MD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, Clinical Neuroscience Research Unit, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Ranganathan M, Cortes-Briones J, Radhakrishnan R, Thurnauer H, Planeta B, Skosnik P, Gao H, Labaree D, Neumeister A, Pittman B, Surti T, Huang Y, Carson RE, D'Souza DC. Reduced Brain Cannabinoid Receptor Availability in Schizophrenia. Biol Psychiatry. 2016 Jun 15;79(12):997-1005. doi: 10.1016/j.biopsych.2015.08.021. Epub 2015 Aug 29. PMID 26432420